CLINICAL TRIAL: NCT05196022
Title: Impact of Treating Unilateral and Bilateral Severe-to-profound Sensorineural Hearing Loss on Productivity and Social Wellbeing
Brief Title: Hear Again, Work Again
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Cochlear (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-0306
Record Dates: First submitted 2021-12-03; First posted 2022-01-19 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-05

CONDITIONS: Hearing Loss, Sensorineural, Severe; Hearing Loss, Sensorineural, Bilateral; Hearing Loss, Unilateral; Hearing Loss, Sensorineural, Profound; Cochlear Implants
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Unilateral | interventions — Cochlear Implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- G1: Patients with bilateral severe to profound hearing loss that would qualify for reimbursement of en cochlear implant but will not opt for a cochlear implant.
- G2: Patients with bilateral severe to profound hearing loss that would qualify for reimbursement of en cochlear implant and receive a cochlear implant
  Interventions: Other: Cochlear implant
- G3: Patients with a single-sided deafness in an acute setting
- G4: Patients with a single-sided deafness in a chronic setting

INTERVENTIONS:
Other: Cochlear implant — G2 will receive a cochlear implant during the study
  Groups: G2

SUMMARY:
Project synopsis:

This prospective cohort study investigates impact of (1) hearing loss and (2) cochlear implantation on cost and health state on one hand, and employment, productivity and social wellbeing on the other hand in a professionally active group using validated questionnaires.

Participants:

The investigators aim to include 100 professional active adults between 18 and 65 years old. All participants have a bilateral severe-to-profound sensorineural or mixed hearing loss. Due to several reasons such as an optimal hearing aid fitting, the presence of a residual hearing or physical contra-indications, half of these participants will not be implanted with CI. Additionally, 100 participants with a single-sides deafness (SSD) in the acute or chronic setting (SDD present for at least three months) will be included.

Study design

Study measures:

All audiological tests and patient-reported outcome measures will be included in this test protocol and repeated throughout the follow-up visits depending on aided or unaided setting. The cognitive evaluation will be executed during the first and last test moment.

The investigators anticipate that the protocol will take 1 hour per follow-up in the hospital (audiological testing and to go over the questionnaires), plus an extra hour at home to fill out the questionnaires. For the cognitive tests, an extra hour in the hospital will be scheduled.

Hypothesis

As a primary endpoint, the investigators anticipate demonstrating that severe-to-profound hearing loss has a significant impact on sick leave and self-reported productivity.

Health state will also be analyzed as a secondary endpoint because the investigators anticipate only marginal improvement (if any) on these instruments due to the lack of sensitivity and responsiveness, even in this population. The investigators will also determine the rate of usage and non-usage at this long-term follow-up to demonstrate the utility of cochlear implants.

Statistical analysis

IBM SPSS Statistics (IBM; Armonk, NY) will be used for the statistical analyses. The participants' hearing profiles will be summarized using descriptive statistics (median, and range). In view of the sample size, non-parametric tests and linear mixed models (to describe evolution in time and difference between groups) will be used. Quantitative data will be presented as median and range (minimum and maximum). Descriptives will be used to summarize the outcomes of the subjective data logging. For the speech perception in noise results, a Wilcoxon signed-rank test will be used. In addition, to correct for the multiple speech in noise test configurations, Holm's correction will be applied. The level of significance will be set at p.0.05.

Data storage

REDCap (Research Electronic Data Capture) is a secure, web-based application designed exclusively to support data capture for research studies. REDCap provides an interface for data entry (with data validation) and audit trails for tracking data manipulation and export procedures. Data will be pseudomized before storage in REDCap.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Unilateral or bilateral severe-to-profound sensorineural or mixed hearing loss
* Ability to understand and speak Dutch
* Resident in Flanders

Exclusion Criteria:

* Already implanted with a cochlear implant
* Conductive hearing loss
* Congenital hearing loss
* Inability to complete audiological or cognitive evaluation
* Inability to complete questionnaires

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators aim to include patients with severe-to-profound hearing loss that would qualify for reimbursement of a cochlear implant (CI) (G1 + G2). A proportion of these patients will not opt for CI (e.g. because of optimal hearing aid fitting) and will be included as G1. Patients receiving CI are G2. In addition, the investigators aim to include 50 single-sided deafness in the acute setting (G3) and 50 single-sided deaf patients (G4).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Change in sick leave after 3, 6 and 12 months | Baseline; 3 months; 6 months; 12 months
  Work Productivity and Activity Impairment Questionnaire - Specific Health Problem. To determine the impact of hearing loss on work productivity the investigators will use "hearing loss" as the specific health problem to develop the WPAI: Hearing as a responsive tool to evaluate work productivity in a hearing impaired population. This questionnaire consists of six items. Four different outcomes will be calculated: percent work time missed due to health, percent impairment while working due to health, percent overall work impairment due to health and percent activity impairment due to health. A higher percentage (minimum=0%; maximum= 100%) on each subscale indicates a greater impact on work productivity.
Change in self-reported productivity after 3, 6 and 12 months | Baseline; 3 months; 6 months; 12 months
  The Work Limitations Questionnaire (WLQ) measures the degree to which employed individuals are experiencing limitations on-the-job due to their health problems, and health-related productivity loss (Presenteeism). The WLQ items ask respondents to rate their level of difficulty or ability to perform specific job demands. The WLQ's 25 items are aggregated into four scales: time management scale, physical demands scale, cognitive job tasks and output demands scale. Scale score range from 0 (limited none of the time) to 100 (limited all of the time) and represent the reported amount of time in the prior two weeks respondents were limited on-the-job. Additionally, using an algorithm, WLQ scale scores can be converted into an estimate of productivity loss where a high score indicates that the participant is limited for a great amount of time.

SECONDARY OUTCOMES:
Change in health state based on the EQ-5D-5L after 3, 6 and 12 months | Baseline; 3 months; 6 months; 12 months
  The EQ-5D-5L is a descriptive system to evaluate the health state and consists of five dimensions: mobility, self-care, usual activities, pain/discomfort, anxiety/depression with five response alternatives each. Based on these responses an EQ-5D-5L profile can be obtained with an index value between 0 (death) and 1 (perfect health). A visual analogue scale with a scale from 0 (worst possible health status) to 100 (best possible health status) is included to assess the self-perceived health.
Change in health state based on the Health Utilities questionnaire (HUI-3) after 3, 6 and 12 months | Baseline; 3 months; 6 months; 12 months
  The HUI-3 is a seventeen-item questionnaire measuring QoL and health states. HUI-3 can be applied in a wide variety of subjects, diseases, interventions and therapies. The following three different types of outcome measures can be derived: attribute levels, single- and multi-attribute scores. Attribute levels represent health states and are as follows: vision, hearing, speech, emotion, pain, ambulation, dexterity and cognition. Levels range from one (no disability) to seven (severe disability). Single-and multi attribute scores are derived from these attribute levels and range from 0 (dead) to 1 (perfect health). Single-attribute scores represent Health Related Quality of Life (HRQoL) per attribute level, while multi-attribute scores provide a general HRQoL value.
Subjective data logging CI | 3 months
  The amount of hours a day and days a week the CI is used.
Objective data logging CI | 3 months
  The amount of hours a day and days a week the CI is used.
Subjective data logging CI | 6 months
  The amount of hours a day and days a week the CI is used.
Objective data logging CI | 6 months
  The amount of hours a day and days a week the CI is used.
Subjective data logging CI | 12 months
  The amount of hours a day and days a week the CI is used.
Objective data logging CI | 12 months
  The amount of hours a day and days a week the CI is used.
Change in treatment-specific health-related Quality of Life based on the Nijmegen Cochlear Implant Questionnaire (NCIQ) after 3, 6 and 12 months | Baseline; 3 months; 6 months; 12 months
  The NCIQ assesses the health-related states on psychological, physical and social domain in CI users based on 60-items formulated as statements. Those items are divided into six subdomains: basic sound perception, advanced sound perception, speech production, self-esteem, activity and social interaction. For every statement, except the last five statements, never (1 point), sometimes (2 point), often (3 points), mostly (4 points) and always (5 points) are possible response alternatives. The last five items represent the ability to perform a stated task. The following response alternatives are possible: no (1 point), poorly (2 points), moderate (3 points), adequate (4 points) and good (5 points). When the item is not applicable for the participants, the item can be marked as 'not applicable'. For every subdomain, the percentage can be calculated. A lower score indicates a poorer quality of life.
Change in treatment-specific health-related Quality of Life based on the Amsterdam Inventory for Auditory Disability and Handicap (AIADH) after 3, 6 and 12 months | Baseline; 3 months; 6 months; 12 months
  The AIADH is a 30- item self-reported questionnaire to assess self-reported disability in everyday hearing. The response scale for each item is a four-point Likert scale measuring how often the respondent is able to hear effectively in a specific situation (0 = almost always, 1 = frequently, 2 = occasionally, or 3 =almost never). Higher scores denote higher impairment.
Change in general sense of preceived self-efficacy after 3, 6 and 12 months | Baseline; 3 months; 6 months; 12 months
  The General Self-Efficacy Scale (GSE) was created to assess a general sense of perceived self-efficacy with the aim in mind to predict coping with daily hassles as well as adaptation after experiencing all kinds of stressful life events. The responses to the 10 items are made on a four-point scale, resulting in a final composite score with a range from 10 to 40. A higher score on the GSE indicates more self-efficacy.
Change in medical cost after 3, 6 and 12 months | Baseline; 3 months; 6 months; 12 months
  The iMTA Medical Consumption Questionnaire (iMCQ) is a generic instrument for measuring medical costs. It includes 18 questions related to frequently occurring contacts with health care providers. The costs for each type of health care provider (i.e. primary, secondary, psychosocial, occupational, and complementary care) will be calculated as the sum of the amount of each resource used, multiplied by its associated unit costs. Costs for overall health care use as well as costs for health care use without hearing related contacts will be calculated, similar to Nachtegaal J, et al. Int J Audiol. 2010. Tariffs will be used as reported by the Belgian National Institute for Health and Disability Insurance (RIZIV-INAMI).
Change in anxiety and depression after 3, 6 and 12 months | Baseline; 3 months; 6 months; 12 months
  The Hospital Anxiety and Depression Scale (HADS) assesses anxiety and depressive symptoms and consists of fourteen statements respondents need to answer based on the degree to which the statement is true. Four response alternatives are given per statement, each corresponding with a score ranging from zero to three. The questionnaire is divided into two subscales; anxiety and depression, each comprising seven questions. Scores are calculated per subscale and range from 0 to 21. A score of zero to seven is considered normal, whereas scores of eleven or higher indicate presence of a mood disorder and scores ranging from eight to ten suggest a mood disorder could be present (borderline).
Change in need for recovery after work after 3, 6 and 12 months | Baseline; 3 months; 6 months; 12 months
  Need for recovery after work will be measured using the need for recovery scale, an six-item scale assessing the short-term effects of fatigue caused by work activities. It is a subscale of the Dutch questionnaire on the experience and assessment of work (VBBA, Vragenlijst Beleving en Beoordeling van de Arbeid). Four response alternatives are possible for each item: always (3 points), often (2 points), sometimes (1 point) and never (0 points). The total score on this subscale is between 0 and 18. A higher score indicates a higher need for recovery after work.
Change in socio-professional reintegration after 3, 6 and 12 months | Baseline; 3 months; 6 months; 12 months
  The Quickscan will be conducted in participants who are on sick leave. Based on 18 items with a six-point Likert scale from zero to five the need for guidance to improve the socio-professional reintegration can be identified. A higher score indicated a higher need for guidance.
Change in cognition based on the Repeatable Battery for the Assessment of Neuropsychological Status for Hearing impaired individuals (RBANS-H) after 3, 6 and 12 months | Baseline; 12 months
  The RBANS-H is a comprehensive cognitive test battery. The oral instructions and auditory stimuli of the RBANS are supported by written explanations and visual stimuli in the RBANS-H, which makes the RBANS-H usable for assessing patients with hearing loss. Five cognitive domains, i.e. immediate memory, visuospatial/ constructional, language, attention and delayed memory will be assessed with the RBANS-H using twelve subtests. The raw score for each subtest will be converted to norm scores using age-specific index score tables. Those index scores will be added up to obtain the total scale score of cognition which is convertible to an age-corrected standard score with a mean of 100 and a standard deviation of 15.
Change in visuospatial short-memory after 3, 6 and 12 months | Baseline; 12 months
  The Corsi Block-Tapping task will be used to evaluate the visuospatial short-term memory. During this test, nine blocks are presented on a computer screen where a sequence of blocks will light up. The participant has to designate the correct blocks in the correct order. Two different sequences of each block will be presented starting with two items for each sequence. When the participant can reproduce one of the two sequence correctly, one item will be added to the sequence. When the participant is not able to repeat either sequence the test ends. The amount of blocks in the last correct sequence will be the corsi span score. A higher score indicates a better visuospatial short-term memory.
Change in hearing thresholds after 3, 6 and 12 months | Baseline; 3 months; 6 months; 12 months
  The pure tone audiometry will be performed in a soundproof booth using insert-earphones, a bone conductor and a two-channel AC-40 audiometer (Interacoustics, Assens, Denmark). The modified Hughson-Westlake technique will be used to investigate the air conduction (AC) ear specific thresholds at 125 Hz, 250 Hz, 500 Hz, 1000 Hz, 2000 Hz, 3000 Hz, 40000 Hz, 6000 Hz and 8000 Hz and bone conduction (BC) ear specific thresholds at 250 Hz, 500 Hz, 1000 Hz, 2000 Hz, 3000 Hz and 40000 Hz when the AC thresholds between 250 and 4000 Hz exceed normality levels (20 decibel hearing level (dBHL)). Afterwards, an unaided and best aided free field measurement will be conducted with the loudspeaker at 0° azimuth and a distance of 1 meter from the participant.
Change in speech perception in quiet after 3, 6 and 12 months | Baseline; 3 months; 6 months; 12 months
  To investigate speech comprehension in quiet the Dutch NVA lists from the Dutch Society for Audiology (Nederlandse Vereniging voor Audiologen) will be executed. The list that consists of ten monosyllabic words composed of a consonant-vowel-consonant and one training word will be presented at 65 dBHL. Both a free field unaided and best aided measurement will be executed where the participant will be placed at 0° azimuth at 1 meter distance of the loudspeaker.
Change in speech perception in noise after 3, 6 and 12 months | Baseline; 3 months; 6 months; 12 months
  To evaluate the speech comprehension in noise an adaptive procedure by the Leuven Intelligibility Sentences Test will be executed in free field in two test conditions (unaided and best aided). One list of this SPIN-test contains 10 sentences. The same test set-up as the speech perception in quiet test will be used. For every test condition- the speech reception threshold (SRT) will be calculated as the average speech level of the last five sentences and the imaginary 11th sentence.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Van Rompaey, Study Director — University Hospital, Antwerp
Locations (1):
- Universitair Ziekenhuis Antwerpen, Edegem, Antwerpen, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Philips C, Jacquemin L, Lammers MJ, Wouters K, Moyaert J, Vanderveken O, Van Rompaey V. Impact of hearing impairment and cochlear implantation on productivity and social well-being in a professionally active but severely hearing-impaired group: protocol of the 'Hear again, work again' longitudinal prospective cohort study. BMJ Open. 2023 Mar 8;13(3):e064514. doi: 10.1136/bmjopen-2022-064514. PMID 36889821